CLINICAL TRIAL: NCT04617808
Title: Predictive Score for Non-traumatic Secondary Headache After an Emergency Call
Acronym: CEPHAREG
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Régional d'Orléans (Other)
Responsible Party: Sponsor
Other Study IDs: CHRO-2019-02
Record Dates: First submitted 2020-10-28; First posted 2020-11-05 (Actual); Last update posted 2022-03-28 (Actual); Status verified 2022-03

CONDITIONS: Headache; Emergencies
Keywords: headache; Emergency
MeSH Terms: conditions — Headache; Emergencies | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Headache pattern: Telephone call from center 15 for the headache pattern
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — The regulatory scheme applied to all investigative centers is as follows:
  * Call from Center 15 by a major patient for secondary headache no traumatic. (i.e. not having been the victim of a head trauma during the 48 hours preceding the call)
  * Detection of the pattern of "non-traumatic headache", by the regulatory assistant medical with registration of the word "cephareg" in the medical regulation software in order to alert the regulator about the possible inclusion of the patient
  * If possible, patient information on the collection of their data for research and possibility of opposing
  * Filling of a medical questionnaire by the regulating doctor
  * Weekly collection of medical questionnaires by investigating doctors

SUMMARY:
The study objective was to identify predictive criteria of severe non-traumatic secondary headache among the information gathered during telephone interview conducted by the on-call regulating physician at the Centre15.

DETAILED DESCRIPTION:
Headache accounted for 1% of outpatient consultations, 2% of hospital emergency department visits and, at the French national level, 1% of complaints motivating calls to the prehospital emergency medical service units (The French, physician-led Emergency Calls Centers , called either "Center 15" or Service d'Aide Médicale d'Urgence [SAMU]). In 2009, the French "SAMU-Urgences de France" society proposed a classification and diagnostic tool for evaluating the headache patient, which is yet to be validated by a clinical study. Most patients with headache spontaneously consulted the emergency department (ED) and only 4 to 5% of patients entered ED through ambulance, fire and rescue department, medicalized ambulance (SMUR), or police. Patients attending emergency service for unusual sudden headache arriving by ambulance had a higher frequency of subarachnoid haemorrhage.

Headache studies have mainly been conducted in the ED. The Ottawa rule published by Perry et al. in 2013 proposed criteria for conducting explorations for subarachnoid hemorrhage (SAH) in patients over 15 years of age with severe, non-traumatic headache, having reached maximum intensity within one hour.

Unlike the primary headaches, secondary headaches are associated with underlying causes. Among the severe secondary headaches (SSH) (4 to 5% of headaches), non-traumatic subarachnoid haemorrhage was not diagnosed in 5.4% to 12% of cases in ED resulting in increase in mortality from 5 to 14%.

In 2018, French guidelines for the emergency management of headache recognized criteria likely to be at risk of Severe Secondary Headache, requiring explorations in emergencies for sudden headaches or thunderclaps headaches (i.e. reaching maximum intensity in less than a minute), recent headaches or progressive worsening (<7 days) and unusual, association with fever (apart from an obvious cause), association with signs of neurological impairment, suspicion of carbon monoxide poisoning, immunosuppression (neoplasia, HIV). Any unusual headache in a patient with recurrent paroxysmal or chronic headache should be considered secondary until proven otherwise. Subarachnoid hemorrhages were present in 11% of patients with sudden, intense and unusual headache.

In the French department of Loiret, patients with subarachnoid haemorrhage required a transfer out of the department to the nearest regional referral teaching hospital, by lack of adequate equipment and expertise for interventional neurology. Early diagnosis was therefore critical. In fact, an untreated cerebral aneurysm rupture increased bleeding recurrence by 3-4% in the first 24 hours.

ELIGIBILITY:
Inclusion Criteria:

* Telephone call from center 15 for the headache pattern
* Age ≥ 18
* Non-opposition expressed by the patient
* Or non-opposition delayed (adults with cognitive disorders, protected adults, clinical situations judged to be serious by the Medical Regulation Assistant, physician regulator, incoming call flow, call by close or trusted person)

Exclusion Criteria:

* Head trauma < 48 hours
* Moribund patient
* Non-affiliation to a social security scheme
* Opposition to the continuation of the study expressed orally by the patient or by return mail within 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients presenting all the inclusion criteria and not showing any of the non-inclusion criteria will be included prospectively and consecutively when calling for medical regulation from the SAMU 45. The patients will be included in the study by the doctor regulator.
Sampling Method: Non-Probability Sample
Enrollment: 715 (Actual)
Dates: Start 2020-10-21 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with diagnosis of non-traumatic secondary headache | Day 21
  Proportion of patients with diagnosis of non-traumatic secondary headache attended by the French emergency services operating

SECONDARY OUTCOMES:
Proportion of patients requiring an admission to Intensive Care Unit | Day 2
  Proportion of patients requiring an admission to the Intensive Care Unit between triage in the emergency department (Day 0) and Day 2
Number of patients with early mortality | Day 7
  Number of patients who died in hospital at day 7

CONTACTS AND LOCATIONS:
Overall Officials: JULIEN PASSERIEUX, Dr, Study Chair — CHR ORLEANS
Locations (2):
- France (2):
  - Regional Hospital center of Orleans, Orléans
  - CHRU de Tours, Tours

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Burch RC, Loder S, Loder E, Smitherman TA. The prevalence and burden of migraine and severe headache in the United States: updated statistics from government health surveillance studies. Headache. 2015 Jan;55(1):21-34. doi: 10.1111/head.12482. Erratum In: Headache. 2015 Feb;55(2):356. PMID 25600719
- [Background] Goldstein JN, Camargo CA Jr, Pelletier AJ, Edlow JA. Headache in United States emergency departments: demographics, work-up and frequency of pathological diagnoses. Cephalalgia. 2006 Jun;26(6):684-90. doi: 10.1111/j.1468-2982.2006.01093.x. PMID 16686907
- [Background] Valade D. The Emergency Headache Center at the Lariboisiere Hospital: 7 years with more than 70,000 patients. Intern Emerg Med. 2008 Oct;3 Suppl 1:S3-7. doi: 10.1007/s11739-008-0191-6. PMID 18785014
- [Background] Perry JJ, Sivilotti MLA, Sutherland J, Hohl CM, Emond M, Calder LA, Vaillancourt C, Thirganasambandamoorthy V, Lesiuk H, Wells GA, Stiell IG. Validation of the Ottawa Subarachnoid Hemorrhage Rule in patients with acute headache. CMAJ. 2017 Nov 13;189(45):E1379-E1385. doi: 10.1503/cmaj.170072. PMID 29133539
- [Background] Perry JJ, Stiell IG, Sivilotti ML, Bullard MJ, Hohl CM, Sutherland J, Emond M, Worster A, Lee JS, Mackey D, Pauls M, Lesiuk H, Symington C, Wells GA. Clinical decision rules to rule out subarachnoid hemorrhage for acute headache. JAMA. 2013 Sep 25;310(12):1248-55. doi: 10.1001/jama.2013.278018. PMID 24065011
- [Background] Pari E, Rinaldi F, Gipponi S, Venturelli E, Liberini P, Rao R, Padovani A. Management of headache disorders in the Emergency Department setting. Neurol Sci. 2015 Jul;36(7):1153-60. doi: 10.1007/s10072-015-2148-7. Epub 2015 Mar 10. PMID 25754613
- [Background] Chey WY, Kusakcioglu O, Dinoso V, Lorber SH. Gastric secretion in patients with chronic pancreatitis and in chronic alcoholics. Arch Intern Med. 1968 Nov;122(5):399-403. No abstract available. PMID 5687926